CLINICAL TRIAL: NCT04742959
Title: A Phase Ib/II, Multicenter, Open-Label Study of TT-00420 Tablet, as Monotherapy or in Combination Regimens, in Patients With Advanced Solid Tumors
Brief Title: Study of TT-00420 (Tinengotinib) Tablet as Monotherapy and Combination Therapy in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT420X1103
Expanded Access: NCT06370013 (Available)
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor; Cholangiocarcinoma; HER2-negative Breast Cancer; Triple Negative Breast Cancer; Bladder Cancer; Small-cell Lung Cancer; Prostate Cancer; Thyroid Cancer; Sarcoma; Gastric Cancer; Gallbladder Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Triple Negative Breast Neoplasms; Urinary Bladder Neoplasms; Small Cell Lung Carcinoma; Prostatic Neoplasms; Thyroid Neoplasms; Sarcoma; Stomach Neoplasms; Gallbladder Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Study will consist of three arms: Arm A (TT-00420 Tablet Monotherapy), Arm B (TT-00420 tablet in combination with nab-paclitaxel (Abraxane®)) and Arm C (PK Run-in Study of TT-00420 Tablet).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy Cohorts (Experimental): TT-00420 tablets will be administered once daily in 28-day cycles.
  Interventions: Drug: TT-00420
- Dose Escalation Cohorts (Combination Therapy) (Experimental): TT-00420 tablets will be administered once daily in 28-day cycles. Nab-paclitaxel 100 mg/m^2 will be administered intravenously on Day 1, 8, and 15 of each 28-day cycle. Dose escalation will be guided by a 3+3 design in Phase Ib to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: TT-00420; Combination Product: Nab-Paclitaxel
- PK Run-in Cohorts (Experimental): TT-00420 tablets will be administered once or twice daily in 28-day cycles according to assigned cohort.
  Interventions: Drug: TT-00420

INTERVENTIONS:
Drug: TT-00420 — TT-00420 tablet will be administered orally once daily per protocol defined schedule.
Combination Product: Nab-Paclitaxel — Nab-Paclitaxel would be administered via infusion on Day 1,8, and 15 of 28-day cycle
  Arms: Dose Escalation Cohorts (Combination Therapy)

SUMMARY:
This is a Phase Ib/II, multicenter, open-label study to evaluate the safety and preliminary efficacy of TT-00420 tablet, as monotherapy or in combination regimens, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Study consists of three arms, Arm A is a Phase Ib/II study of TT-00420 tablet monotherapy, Arm B is a Phase Ib/II study of TT-00420 tablet in combination with nab-paclitaxel (Abraxane®) and Arm C is a PK run-in study of TT-00420 tablet.

Arm A: TT-00420 Tablet Monotherapy Phase Ib will enroll patients with preferred indications including metastatic cholangiocarcinoma, HER2-negative breast cancer including TNBC, bladder cancer, small cell lung cancer, prostate cancer, thyroid cancer, sarcoma, gastric cancer, gallbladder cancer and other advanced solid tumors to receive TT-00420 monotherapy. Based on preliminary efficacy results, Phase II will enroll additional patients in select indications to evaluate the efficacy of TT-00420 monotherapy.

Arm B: TT-00420 tablet in combination with nab-paclitaxel (Abraxane®) Arm B will enroll patients with metastatic HER2-negative breast cancers, including triple-negative breast cancer (TNBC). Phase Ib will be a dose escalation study of TT-00420 in combination with nab-paclitaxel, guided by 3+3 design, to determine a Recommended Phase 2 Dose (RP2D). Phase II will enroll additional patients with metastatic HER2-negative breast cancers to further evaluate the efficacy of the combination regimen.

Arm C: PK Run-in Study of TT-00420 Tablet Arm C will enroll patients with preferred indications including cholangiocarcinoma, TNBC/HER2- negative breast cancer, prostate cancer, sarcoma, hepatocellular carcinoma (HCC), bladder cancer, small cell lung cancer, thyroid cancer, gastric cancer, gallbladder cancer and other advanced solid tumors to receive TT-00420 monotherapy administered as once daily (q.d.) or twice daily (b.i.d.).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Histopathological or cytologically documented locally advanced or metastatic solid tumors who have no available standard therapeutic treatment options
3. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Adequate organ function confirmed at screening and within 10 days of initiating treatment, as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Hemoglobin (Hgb) ≥ 8 g/dl
   * Platelets (plt) ≥ 75 x 10^9/L
   * AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 x ULN
   * Calculated creatinine clearance ≥ 50 mL/min (Cockcroft Gault formula)
6. Negative pregnancy test within 72 hours before starting study treatment in all premenopausal women and women < 12 months after the onset of menopause
7. Must agree to take sufficient contraceptive methods to avoid pregnancy during the study and until at least 6 months after ceasing study treatment
8. Able to sign informed consent and comply with the protocol

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control
3. Patients with any hematologic malignancy, including leukemia (any form), lymphoma, and multiple myeloma
4. Patients with a history of primary central nervous system tumors or carcinomatous meningitis.
5. Patients with the following mood disorders as judged by the Investigator or a psychiatrist:

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia; a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
   * ≥ CTCAE grade 3 anxiety
6. Impaired cardiac function or significant diseases, including but not limited to any of the following:

   * left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Congenital long QT syndrome
   * QTcF ≥ 480 msec on screening ECG
   * Unstable angina pectoris ≤ 3 months prior to starting study drug
   * Acute myocardial infarction ≤ 3 months prior to starting study drug
7. Patients with:

   * unresolved diarrhea ≥ CTCAE grade 2, or
   * impairment of gastrointestinal (GI) function, or
   * GI disease that may significantly alter the absorption of TT-00420
8. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., uncontrolled hypertension, uncontrolled hypertriglyceridemia, or active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
9. Patients who have received chemotherapy, targeted therapy, or immunotherapy ≤ 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
10. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
11. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
12. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 4 weeks prior to starting study drug.
13. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium or any other coumarin-derivative anticoagulants
14. Patients who have received systemic corticosteroids ≤ 2 weeks prior to starting study drug or who have not recovered from the side effects of such treatment.
15. Patients who are currently receiving treatment with strong CYP3A inhibitors or inducers ≤ 2 weeks prior to starting study drug.
16. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory; patients with well controlled HIV might be enrolled)
17. Known history of active infection with Hepatitis B or Hepatitis C
18. Has received a live-virus vaccination within 30 days of planned first dose
19. Inability to swallow or tolerate oral medication
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's safe participation and compliance in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Up to 30 days from study discontinuation
  As assessed per NCI Common Toxicity Criteria for Adverse Events, version 5.0
Dose limiting toxicity (DLT) | Up to 28 days from the first dose
  Dose escalation cohorts are monitored and assessed using the NCI Common Toxicity Criteria for Adverse Events, version 5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 9 months.
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Disease Control Rate (DCR) | Through study completion, an average of 9 months.
  Defined as CR + PR + stable disease (SD) based on RECIST version 1.1.
Duration of Objective Response (DOR) | Through study completion, an average of 9 months.
  Duration of response for CR or PR based on RECIST version 1.1.
Progression Free Survival (PFS) | From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall Survival (OS) | From first study drug administration until the date of death from any cause, assessed up to 24 months
Area under the curve (AUC0-∞) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)
  Blood samples will be collected at designated time points for pharmacokinetic analysis of TT-00420 and/or nab-paclitaxel.
Area under the curve (AUC0-t) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)
  Blood samples will be collected at designated time points for pharmacokinetic analysis of TT-00420 and/or nab-paclitaxel.
Maximum observed concentration (Cmax) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)
  Blood samples will be collected at designated time points for pharmacokinetic analysis of TT-00420 and/or nab-paclitaxel.
Half-life (T1/2) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)
Time to Maximum Concentration (Tmax) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)
Volume of Distribution (Vd) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 28 days)

OTHER OUTCOMES:
Genetic Alteration Status | Through study completion, an average of 9 months
  Evaluation of biomarkers, including but not limited to, fibroblast growth factor receptor (FGFR) mutation status

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A. Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - The University of Chicago, Chicago, Illinois
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Gabrail Cancer Center Research, Canton, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No